CLINICAL TRIAL: NCT03727152
Title: Maintenance of Switching From Protease Inhibitor/Ritonavir to Generic Single Tablet Regimen of Tenofovir Alafenamide/Emtricitibine/Dolutegravir in Virologically Suppressed HIV-infected Adults
Brief Title: Switching From Protease Inhibitor/Ritonavir to Generic Single Tablet Regimen of Tenofovir Alafenamide/Emtricitibine/Dolutegravir
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Faculty of Medical Sciences, Radboud University of Medical Center (Unknown); Department of Pharmaceutical care, Faculty of Pharmacy, Chiang Mai University (Unknown); Police General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 256
Record Dates: First submitted 2018-10-26; First posted 2018-11-01 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: HIV
Keywords: generic TAF/E/D; virologically suppressed HIV-infected adults; pharmacokinetics (PK) parameters of DTG; psychiatric symptoms; metabolic syndrome; ASCVD risk; liver fibrosis
MeSH Terms: conditions — Metabolic Syndrome; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- generic single tablet regimen of tenofovir alafenamide/e (Other): HIV infected adults currently on protease inhibitor/ritonavir will switch to use generic single tablet regimen of tenofovir alafenamide/emtricitibine/dolutegravir to see if the single tablet can continue to suppress viral replication and be used as a maintenance regimen
  Interventions: Drug: generic single tablet TAF/FTC/DTG

INTERVENTIONS:
Drug: generic single tablet TAF/FTC/DTG — HIV-infected adults who are virologically suppressed and on protease inhibitor/ritonavir are switched to generic single tablet regimen of tenofovir alafenamide/emtricitibine/dolutegravir

SUMMARY:
This is a phase III, multicenter, open-label, single-arm study of 190 virologically suppressed HIV-infected adults

DETAILED DESCRIPTION:
The fundamental principle of regimen switching is to maintain viral suppression without jeopardizing future treatment options. The reasons to consider regimen switching in the viral suppressed population are to simplify the regimen by reducing the pill burden and dosing frequency, to increase the tolerability, reduce the adverse effects as well as long-term toxicities, to prevent drug-to-drug interactions and to avoid the dietary requirements.

Generic TAF/E/D (tenofovir alafenamide 25mg/emtricitabine 200mg/dolutegravir 50 mg), a single-tablet once daily regimen, will be an affordable regimen with the potential characteristics such as reduced pill burden, less drug to drug interaction and toxicities. The generic form (Mylan) is recently received the tentative approval from the U.S. Food and Drug Administration (FDA) under the U.S. President's Emergency Plan for AIDS Relief (PEPFAR). Whether DTG-containing regimen is a better option than protease inhibitors among resource-limited settings during the decisions for second-line treatment options, is needed to be evaluated.

All participants will be switched from their pre-study ART regimen to a single tablet regimen (STR) of TAF/FTC/DTG 25/200/50mg once daily.

ELIGIBILITY:
Inclusion Criteria:

1. Documented HIV-1 infection
2. Aged ≥18 years old
3. Female participant may be eligible to participate if she:

   is of non-childbearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea or >=54 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy, or bilateral oophorectomy or, is of child-bearing potential, with a negative pregnancy test at both Screening and week 0 and agrees to use one of the protocol-defined methods of contraception to avoid pregnancy.
4. On current ART for at least 6 months prior to study entry
5. Current ART includes boosted protease inhibitors
6. No more than one HIV-1 plasma RNA >50 copies/mL and <200 copies/L (only one 'blip') in the past 6 months with a subsequent HIV-1 plasma RNA <50 copies/mL
7. HIV-1 plasma RNA <50 copies/mL at screening visit
8. No prior or current exposure to integrase strand transfer inhibitor (INSTI)
9. Have signed the informed consent form

Exclusion Criteria:

1. Breastfeeding female
2. Pregnancy or positive UPT at screening
3. Calculated creatinine clearance as estimated by Cockcroft-Gault equation (CrCl) <60 mL/min,
4. Alanine aminotransferase (ALT) >2.5 x ULN,
5. Concomitant use of any of the following medications:

(1) aluminum and magnesium-containing antacids, proton-pump inhibitors (2) anticonvulsants: carbamazepine, oxcarbamazepine, phenobarbital, phenytoin (3) antimycobacterials: rifabutin, rifampin, rifapentine (4) St. John's wort

6. Alcohol or drug abuse that, in the opinion of the investigator, would interfere with completion of study procedures

7. Any serious illness that, in the opinion of the investigator, would interfere with completion of study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
number of subjects with undetectable viral load | 48 weeks
  Proportion of participants with plasma HIV-1 RNA <50 copies/mL using Snapshot algorithm at week 48

SECONDARY OUTCOMES:
Proportion of participants without tolerability failure | weeks 24 and weeks 48
  Proportion of participants without tolerability failure
Cmax of DTG | weeks 24 and weeks 48
  maximum plasma concentration (Cmax) of DTG 50 mg
Tmax of DTG | weeks 24 and weeks 48
  time to reach maximal concentration (Tmax) of DTG 50 mg
AUC of DTG | weeks 24 and weeks 48
  area under the curve of a plasma concentration versus time profile (AUC) of DTG 50 mg
T1/2 of DTG | weeks 24 and weeks 48
  elimination half life (T1/2) of DTG 50 mg
Ke of DTG | weeks 24 and weeks 48
  elimination rate constant (Ke) of DTG 50 mg
CL of DTG | weeks 24 and weeks 48
  total plasma clearance (CL) of DTG 50 mg
Anxiety at baseline will be compared to level of anxiety at weeks 24 and weeks 48. | weeks 24 and weeks 48
  Anxiety at baseline will be compared to anxiety level at weeks 24 and weeks 48. Anxiety will be assessed using Hospital Anxiety and Depression Scale (HADS). There are 7 different items that assess the level of anxiety of the participants based on a four-point grading scale specific for each item assessed (i.e., I feel tense or 'wound up'; 0 = not at all; 1 = from time to time, occasionally; 2 = a lot of the time; 3 = most of the time). If the total score is between 0-7, then this is considered to be normal. If the total score is between 8-10, then this is considered borderline abnormal (borderline case). If the total score is between 11-21, then this is considered abnormal (case).
Depression at baseline will be compared to depression level at weeks 24 and weeks 48. | weeks 24 and weeks 48
  Depression at baseline will be compared to depression level at weeks 24 and weeks 48. Depression will be assessed using Hospital Anxiety and Depression Scale (HADS). There are 7 different items that assess the level of depression of the participants based on a four-point grading scale specific for each item assessed (i.e., I still enjoy the things I used to enjoy; 0 = definitely as much; 1 = not quite so much; 2 = only a little; 3 = hardly at all). If the total score is between 0-7, then this is considered to be normal. If the total score is between 8-10, then this is considered borderline abnormal (borderline case). If the total score is between 11-21, then this is considered abnormal (case).
Changes from baseline in fasting lipid profiles | weeks 24 and weeks 48
  Changes from baseline in fasting lipid profiles (HDL, LDL, cholesterol, TG)
Changes from baseline in insulin | weeks 24 and weeks 48
  Changes from baseline in insulin
Changes from baseline in fasting blood glucose levels | weeks 24 and weeks 48
  Changes from baseline in fasting blood glucose levels
Changes from baseline in renal parameters (creatinine, eGFR) | weeks 24 and weeks 48
  Changes from baseline in renal parameters (creatinine, eGFR)
Changes from baseline in transient elastography results | weeks 24 and weeks 48
  Changes from baseline in transient elastography results

CONTACTS AND LOCATIONS:
Overall Officials: Sivaporn Gatechompol, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration
Locations (2):
- Thailand (2):
  - HIV-NAT, Thai Red Cross AIDS Research Centre, Bangkok
  - Police General Hospital, Bangkok